CLINICAL TRIAL: NCT03794206
Title: CD 1009 Rev A Page 1 of 44 23OCT2018 Vesair Balloon Confirmatory Trial (VECTOR) Use of the Next Generation Vesair® Bladder Control System for the Treatment of Stress Urinary Incontinence in Post-Menopausal Women
Brief Title: Vesair Balloon Confirmatory Trial (VECTOR)
Acronym: VECTOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company closure
Sponsor: Solace Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD1009
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Single-arm of subjects who receive treatment with Vesair Balloon
  Interventions: Device: Vesair Balloon

INTERVENTIONS:
Device: Vesair Balloon — Treatment with Vesair Balloon for one year

SUMMARY:
Multicenter, prospective, single-arm study to assess the safety and efficacy of the Vesair Bladder Control treatment in post-menopausal women with Stress Urinary Incontinence (SUI) with follow-up at 1, 3 and 12 months. All subjects will be prospectively treated after the subject has provided informed consent and determination that all study entry criteria have been met.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated with Vesair Balloon within the past 4 years
* Normal voiding function
* Has signed consent
* Willing to undergo cystoscopy
* Available for minimum of 12 months

Exclusion Criteria:

* Last Menstrual Period within past 4 years
* Systemic birth control medication (including implants) or systemic hormone replacement therapy (estrogen or progesterone) in the past 4 years.
* History of urosepsis, bladder infection, urinary tract infection or asymptomatic bacteriuria within the past 3 months.
* Urinary incontinence of neurogenic etiology.
* Prior pelvic surgery that may affect incontinence symptoms (including placement and/or removal of a suburethral sling) within the past 4 years.
* Noninvasive treatment for incontinence, such as nerve stimulation, Botox injections, biofeedback, formal pelvic floor muscle training, and/or vaginal laser therapy, within the past 3 months.
* Taken medications other than anticholinergics that may affect SUI symptoms (such as enobosarm, duloxetine or imipramine) in the past 3 months.
* Taking other pharmacologic agents that may have a significant effect on bladder function unless on the therapy for at least 3 months and intending to continue the same dosage of the medication throughout the trial.
* History of recurrent (>1) kidney stones, or one kidney stone within the past 5 years.
* History of an artificial urinary sphincter.
* Presence of gross hematuria and/or blood clots in the urine.
* History of interstitial or follicular cystitis or other painful bladder syndrome.
* Cystocele verified as Stage 3 or higher by PoP-Q Classification.
* Local genital skin infection.
* Urethral or bladder inflammation and/or edema, or other hypersensitivity to cystoscopy or other urethral manipulations.
* Evidence of involuntary detrusor contractions and/or discomfort during bladder filling up to 300cc.
* Undergoing or anticipating a course of pelvic radiation therapy or with severe pelvic fibrosis from previous radiation therapy.
* Non-ambulatory, bedridden or physically unable to complete test exercises.
* History of recent alcoholism or illicit drug abuse within the last year.
* Immunologically suppressed or immunocompromised.
* History of any neurological disease that could impact bladder function including Parkinson's disease, multiple sclerosis or post-stroke sequelae.
* Uncontrolled diabetes (persistent A1C levels >9 percent).
* History of any malignancy (except non-melanoma skin cancer), unless the cancer was not in the urinary tract, the cancer was stage II or less, the cancer was treated with curative intent, AND there have been no clinical signs or symptoms of the malignancy for at least 2 years.
* Morbid obesity, defined as BMI ≥40.0.
* History of any autoimmune or connective tissue disease or disorder that could impact bladder function

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Provocative Pad Weight | 3 months
  in-office Pad weight test

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rardin, M.D., Principal Investigator — Women and Infants Hospital
Locations (8):
- United States (8):
  - WomanCare, Arlington Heights, Illinois
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology, Hanover, Maryland
  - Chesapeake Urology, Owings Mills, Maryland
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Women and Infants dept of Urogynecology, Providence, Rhode Island
  - Urology of Virginia, Virginia Beach, Virginia
  - Washington Urology, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCammon K, Jacoby K, Kalota S, Snyder J, Cline K, Robertson K, Rardin C, Kahan R, Green L, Zuckerman J, Rovner E. Three-month primary efficacy data for the SUCCESS Trial; a phase III, multi-center, prospective, randomized, controlled study treating female stress urinary incontinence with the vesair intravesical balloon. Neurourol Urodyn. 2018 Jan;37(1):440-448. doi: 10.1002/nau.23324. Epub 2017 Nov 2. PMID 29095516
- See also: Company Website — http://www.solacetx.com